CLINICAL TRIAL: NCT04612842
Title: Engaging Older Adults in Fall Prevention Using Motivational Interviewing (MI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Hiroko Kiyoshi-Teo, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00008993; K23NR018672 (NIH)
Record Dates: First submitted 2020-10-08; First posted 2020-11-03 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Fall; Motivation; Behavior; Coping Behavior
Keywords: Fall prevention; Motivational Interviewing
MeSH Terms: conditions — Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (MI) goup (Experimental): The MI experimental group will receive the same measurements as the control group, and in addition, receive MI-based communication about fall prevention at eight occasions during the 6-month period. MI is an evidence-based communication approach for various health behavior change.
  Interventions: Behavioral: Motivational Interviewing
- Control group (No Intervention): The control group participants will take part in study measurements (self-report and physiologic assessment) for 12-months. Primary assessment measures are at baseline, 6-, and 12-months and will be conducted via phone survey, video assessment, or mail-in calendar.

INTERVENTIONS:
Behavioral: Motivational Interviewing — The PI and two study staff members (interventionists) will conduct study visits and phone calls. The same person will complete participant follow-ups to establish rapport and consistency. All of the study encounters will be audio recorded with participants' permission and study encounter notes will be completed by the interventionist. Interventionists will facilitate MI sessions using the MI guide and a participant handout. The goal of each MI session is to identify a specific fall prevention behavior, the participant's goal with this behavior, readiness to change, specific plan to move toward the goal, barriers and facilitators, and the participant's commitment level to change.
  Arms: Motivational Interviewing (MI) goup

SUMMARY:
This mixed-methods, two-arm, randomized controlled trial will evaluate the impact of Motivational Interviewing (MI) as a follow-up care to patients who received fall prevention recommendations at Oregon Health & Science University Internal Medicine and Geriatrics Clinic provided over 12 months.

DETAILED DESCRIPTION:
The goal of this mixed-methods, two-arm, randomized controlled trial of MI intervention for fall prevention is to evaluate the impact of Motivational Interviewing (MI) as a follow-up care to patients who received fall prevention recommendations at Oregon Health & Science University Internal Medicine and Geriatrics Clinic provided over 12-months. Older adult participants (older than 65) who are at increased risk for falling will be enrolled into the study. Patients will be randomly assigned to two groups: MI and the standard of care group. All participants will have a baseline and 6-months study visit that will include self-report and physiologic assessment. In addition, all participants will receive study measurement phone call at 3-, and 12-months. MI will be provided via video, phone, or in-person one week after the initial visit and then monthly for 6 months. All MI sessions will be recorded and encounter notes will be completed. Purposefully selected participants' MI sessions will be transcribed for qualitative analysis.

ELIGIBILITY:
Inclusion Criteria:

* Oregon Health & Science University (OHSU) Internal Medicine and Geriatrics Clinic patients
* 65 years old or older
* Moderate-to-high risk for falling using the STEADI fall screening and management algorithm
* Cognitively oriented (Mini-Cog≥ 3)
* Able to converse audibly and coherently in English
* Living independently in the community
* Able to receive study phone calls
* Ambulatory with or without assistive device use

Exclusion Criteria:

* Cognitively impaired patients (Mini-Cog< 2)
* Patients who have sensory difficulty with verbal communication (hard-of-hearing despite the use of hearing aids or speech is hard to understand despite a talking device)
* Living in institutions with 24-hour care such as skilled nursing facilities
* Unable to stand without assistance by others
* Life-expectancy of less than 3-months
* Patients participating in other studies that may impact fall-related behavior change

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroko Kiyoshi-Teo, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Interviewing (MI) Group: The MI experimental group will take part in the same study measurements as the control group, and in addition, receive MI-based communication about fall prevention at eight occasions during the 6-month period. MI is an evidence-based communication approach for various health behavior change.
Period: Overall Study
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Started | 101 | 99
Baseline Assessment | 90 | 95
6-month Assessment | 69 | 81
12-month Assessment | 53 | 71
Completed | 53 | 71
Not Completed | 48 | 28
Not completed — Lost to Follow-up | 20 | 11
Not completed — Withdrawal by Subject | 26 | 15
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Motivational Interviewing (MI) Group: The MI experimental group will take part in the same study measurements as the control group, and in addition, receive MI-based communication about fall prevention at eight occasions during the 6-month period. MI is an evidence-based communication approach for various health behavior change.
  Motivational Interviewing: Study interventionists will conduct the remote MI sessions. The same person will complete participant follow-ups to establish rapport and consistency. Study staff will conduct study visits and phone calls. MI sessions will be audio recorded with participants' permission and MI session notes will be completed by the interventionist. Interventionists will facilitate MI sessions using the MI guide and a participant handout. The goal of each MI session is to identify specific fall prevention behaviors, the participant's goals with these behaviors, and promote readiness to change.
- Control Group: The control group participants will take part in study measurements at baseline, 3-, 6-, and 12-months after the benchmark STEADI clinic visit.
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing (MI) Group | Control Group | Total
Number analyzed (Participants) | 90 | 95 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 90 | 95 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.1 (7.6) | 80.9 (7.7) | 80.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 65 | 125
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 85 | 86 | 171
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 90 | 95 | 185
Balance Measure [Mean (Standard Deviation); unit: units on a scale] — Individuals are asked to hold progressively challenging balance position for 10 sections without moving their feet or needing support. The positions are standing with feet side-by-side, semi-tandem (instep of one foot is touching big toe of the other foot), tandem stand (one foot in front of the other- heel touching toe), and stand on one foot. The minimum is 0 and the maximum is 10. A higher number is a better outcome. Population: Some participants were unable to complete the physical function assessments which are secondary measures because of their inability to operate the video call despite study staff's support, or because of infection concerns related to COVID to have a supportive personnel near by (requirement from OHSU IRB).
  units on a scale
    Semi-tandem stand balance: number analyzed (Participants) | 52 | 47 | 99
    Semi-tandem stand balance | 9.96 (0.28) | 9.74 (1.37) | 9.86 (0.97)
    Tandem stand balance: number analyzed (Participants) | 51 | 45 | 96
    Tandem stand balance | 9.33 (1.83) | 8.13 (3.35) | 8.77 (2.7)
    1-legged stand balance: number analyzed (Participants) | 48 | 42 | 90
    1-legged stand balance | 6.71 (3.88) | 5.71 (3.86) | 6.24 (3.88)
    Side-by-side stand balance: number analyzed (Participants) | 52 | 47 | 99
    Side-by-side stand balance | 10 (0) | 9.96 (0.295) | 9.98 (0.20)
Fall Efficacy Scale International- Short [Mean (Standard Deviation); unit: units on a scale] — A 7-item scale widely used to measure levels of concern related to preventing falls while doing certain activities. Individuals self-report their concern from not at all concerned (1) to very concerned (4). Minimum value is 7 and maximum value is 28. Higher FES-I scores is a worse value since it has been positively correlated with decreased activities, future falls, and injury.
  units on a scale | 13.33 (4.46) | 13.83 (5.59) | 13.59 (5.07)
Patient Activation Measure [Mean (Standard Deviation); unit: units on a scale] — A 10-item survey that assesses an individual's knowledge, skills, and confidence to manage one's own health and healthcare. There is an algorithm for scoring on a scale from 0 to 100 that corresponds to one of four levels of patient activation. A score of 0/level 1 is disengaged and overwhelmed and a score of 100/level 4 is maintaining behaviors. A higher score is a better outcome.
  units on a scale | 67.61 (12.86) | 66.69 (13.89) | 67.14 (13.37)
Falls Behavioral Scale [Mean (Standard Deviation); unit: units on a scale] — A list of 30 statements that describes everyday things with a rating from never (1) to always (4) in how often they do each task. The average is taken for a minimum of 0 and maximum of 4. The higher score is a better outcome.
  units on a scale | 3.04 (0.46) | 2.96 (0.46) | 3.00 (0.46)
30-second Sit-to-Stand [Mean (Standard Deviation); unit: units on a scale] — Test leg strength and endurance using a chair with a straight back without arm rests. Individuals are asked to sit in the middle of the chair, place hands on opposite shoulders crossed at the wrists, keep feet flat on the floor, and keep back straight and arms against chest. They are asked to rise to a full standing position and sit back down again for 30 seconds. The number of times an individual comes to a full standing position in 30 seconds is the outcome. Scores range by sex and age-group. For 65-69 year old men, the below average score is under 12 and women is under 11. Higher is better. Population: Some participants were unable to complete the physical function assessments which are secondary measures (4-stage balance test and 30-second sit-to-stand) because of their inability to operate the video call despite study staff's support, or because of infection concerns related to COVID to have a supportive personnel near by (requirement from OHSU IRB).
  units on a scale
    number analyzed (Participants) | 49 | 45 | 94
    (all) | 10 (0.57) | 10.16 (0.6) | 10.1 (4.00)

OUTCOME MEASURES:

1. Primary Outcome: Falls Self-Efficacy Scale-International (FES-I) Results
Description: A 7-item scale, 1-4 self-report rating, widely used to measure levels of concern related to preventing falls. Minimum value is 7 and maximum value is 28. Higher FES-I scores is a worse value since it has been positively correlated with decreased activities, future falls, and injury.
Time Frame: 3-, 6-, and 12-months
Population: We used mixed-effect modeling to measure changes over time, which includes all participants who have outcome measure in at least one time-point. Thus, the analytic sample in the table below looks different from participant flow data. We conducted intent-to-treat analysis (including participants regardless of drop out. No list-wise deletion.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 88 | 94
units on a scale
  3-months | 13.07 (0.57) | 13.71 (0.54)
  6-months | 13.41 (0.59) | 14.35 (0.56)
  12-months | 13.01 (0.67) | 13.82 (0.53)
Statistical Analysis 1: Comparison: Motivational Interviewing (MI) Group vs Control Group; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Fall Behavioral (FAB) Scale Results
Description: A 24-item, 1-4 self-report rating to measure frequency of protective strategies to prevent falling and risky behaviors that facilitate a fall. The average value is calculated with a minimum value of 1 and maximum value of 4. Higher FAB score is a better value since it indicates more consistent fall protective behaviors.
Time Frame: 3-, 6-, and 12-months
Population: We used mixed-effect modeling to measure changes over time, which includes all participants who have outcome measure in at least one time-point. Thus, the analytic sample in the table below looks different from the participant flow data. We conducted intent-to-treat analysis (including participants regardless of drop out. No list-wise deletion.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 90 | 93
units on a scale
  3-months | 3.16 (0.05) | 3.08 (0.05)
  6-months | 3.23 (0.05) | 3.11 (0.05)
  12-months | 3.17 (0.05) | 3.14 (0.05)

3. Secondary Outcome: Patient Activation Measure Results
Description: 100-point, quantifiable scale determining patient engagement in healthcare. Minimum value is 0 and the maximum value is 100. Higher value is a better value since it is indicative of participant's activation with their healthcare.
Time Frame: 3-, 6-, and 12-months
Population: We used mixed-effect modeling to measure changes over time, which includes all participants who have outcome measure in at least one time-point. Thus, the analytic sample in the table below differs from participant flow data. We conducted intent-to-treat analysis (including participants regardless of drop out. No list-wise deletion.)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 90 | 95
score on a scale
  3-months | 70.6 (1.5) | 71.59 (1.44)
  6-months | 70.23 (1.52) | 67.33 (1.45)
  12-months | 70.44 (1.83) | 68.21 (1.63)

4. Secondary Outcome: Level of Confidence to Prevent Falls
Description: 1-item 10-point scale response. Often used in motivational interviewing sessions to gauge an individual's readiness to engage in certain health behaviors. Higher levels of confidence are known to be associated with an increased rate of behavior change.
Time Frame: 3-, 6-, and 12-months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 90 | 95
units on a scale
  3-months | 8.09 (0.18) | 7.74 (0.17)
  6-months | 8.04 (0.18) | 7.79 (0.17)
  12-months | 7.56 (0.24) | 7.67 (0.21)

5. Secondary Outcome: Level of Importance to Prevent Falls
Description: 1-item 10-point scale response. Often used in motivational interviewing sessions to gauge an individual's readiness to engage in certain health behaviors. Higher levels of importance are known to be associated with an increased rate of behavior change.
Time Frame: 3-, 6-, and 12-months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 90 | 95
units on a scale
  3-months | 9.68 (0.12) | 9.41 (0.11)
  6-months | 9.62 (0.12) | 9.63 (0.10)
  12-months | 9.60 (0.12) | 9.59 (0.11)

6. Secondary Outcome: Balance Measure (Feet Side by Side)
Description: Duration that participants can hold feet side-by-side stand (heel to toe standing positions) will be measured up to 10 seconds. Minimum value is 0 seconds and maximum score is 10 seconds. Higher value is a better value since it is indicative of participants' ability to hold balance.
Time Frame: 6- months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: seconds
Groups:
- Motivational Interviewing (MI) Group: The MI experimental group will take part in the same study measurements as the control group, and in addition, receive MI-based communication about fall prevention at eight occasions within 6-months. MI is an evidence-based communication approach for various health behavior change.
  Motivational Interviewing: Study interventionists will conduct the remote MI sessions. The same person will complete participant follow-ups to establish rapport and consistency. Study staff will conduct study visits and phone calls. MI sessions will be audio recorded with participants' permission and MI session notes will be completed by the interventionist. Interventionists will facilitate MI sessions using the MI guide and a participant handout. The goal of each MI session is to identify specific fall prevention behaviors, the participant's goals with these behaviors, and promote readiness to change.
- Control Group: The control group participants will take part in study measurements and routine clinical care.
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 52 | 47
seconds | 10 (0) | 10 (0)

7. Secondary Outcome: Balance Measure (Semi-tandem Stand)
Description: Duration that participants can hold semi-tandem stand (heel to toe standing positions) will be measured up to 10 seconds. Minimum value is 0 seconds and maximum score is 10 seconds. Higher value is a better value since it is indicative of participants' ability to hold balance.
Time Frame: 6- months
Population: The number analyzed differed by time point because of the loss to follow-up and participant withdrawal as indicated in the participant flow data, and participants' willingness and ability to participate in the measurements.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 52 | 47
seconds | 10 (0.17) | 9.79 (0.15)

8. Secondary Outcome: Balance Measure (Tandem Stand)
Description: Individuals are asked to hold a tandem stand (one foot in front of the other- heel touching toe). The minimum is 0 and the maximum is 10. A higher number is a better outcome.
Time Frame: 6-months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 52 | 46
units on a scale | 8.46 (0.56) | 7.47 (0.55)

9. Secondary Outcome: Balance Measure (One-leg Stand)
Description: Individuals are asked to hold a balance position for 10 sections without moving their feet or needing support. This position require standing on one foot. The minimum is 0 and the maximum is 10. A higher number is a better outcome.
Time Frame: 6- months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 50 | 44
seconds | 6.84 (0.68) | 5.28 (0.67)

10. Secondary Outcome: 30-second Sit-to-stand Assessment
Description: Instances that participants can stand from a sitting position will be measured. Minimum value is 0 times. Higher value is a better value since it is indicative of participants' ability to sit-to-stand.
Time Frame: 6-months
Population: Some participants were unable to complete the physical assessment due to physical limitations, access to a video platform, or a support person.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 49 | 45
units on a scale | 11.01 (0.64) | 9.5 (0.61)

11. Secondary Outcome: Number of Participants With Self-reported Falls
Description: Individuals were asked to mail-in reports of falls every month. Participants reporting a fall at least once are counted as a faller. Minimum value is 0. Higher value is worse value as it is indicative that there were more participants who fell during the year.
Time Frame: 1-year
Population: One participant in the MI group had an unreliable reporting of falls due to his unstable memory (ID 1277). Based on the discussion with the Safety Monitoring Council, his data was considered an outlier and removed from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing (MI) Group | Control Group
Number analyzed (Participants) | 90 | 95
Participants | 56 | 50

ADVERSE EVENTS:
Time Frame: 12-months
Description: Fall data were collected systematically via monthly fall calendar. Other adverse events were collected in non-systematic, opportunistic ways.
Arm/Group | Motivational Interviewing (MI) Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/101 | 2/99
Serious Adverse Events (participants affected / at risk) | 11/101 | 13/99
Other Adverse Events (participants affected / at risk) | 54/101 | 62/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Interviewing (MI) Group (N=101) | Control Group (N=99)
Falls (major) (Injury, poisoning and procedural complications) | 3 (3) | 7 (7) — Falls (major): Falls that result in hospitalization.
Death (Metabolism and nutrition disorders) | 2 (2) | 2 (2) — Death
Hip surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hip Surgery
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (2) — Orthostatic hypotension
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Inguinal hernia
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary tract infection
Heart surgery (Vascular disorders) | 0 (0) | 1 (1) — Heart surgery
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Bowel obstruction
Skiing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Skiing injury
Neurosurgery (Nervous system disorders) | 1 (1) | 0 (0) — Neurosurgery
COVID (Infections and infestations) | 1 (1) | 0 (0) — COVID
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Deep vein thrombosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Interviewing (MI) Group (N=101) | Control Group (N=99)
Falls (Injury, poisoning and procedural complications) | 49 (134) | 56 (155) — Falls
Car/bike accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Car/bike accident
Shunt (Eye disorders) | 0 (0) | 1 (1) — Shunt in right eye
Hammer toe (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Hammer toe
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — R Leg pain
Bladder infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Bladder infection
Gut pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gut pain
Cancer removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Cancer removal
Rotator cuff surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Rotator cuff surgery
Nose surgery (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Nose surgery
Headaches (Nervous system disorders) | 1 (1) | 0 (0) — Headaches

LIMITATIONS AND CAVEATS:
Study enrollment & data collection were conducted during the COVID-19 pandemic in Oregon.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT04612842/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT04612842/ICF_001.pdf